CLINICAL TRIAL: NCT06768619
Title: A Multicenter, Randomized, Open-label, Two-formulation, Two-sequence, Two-period Crossover Study to Evaluate the Bioequivalence of Eltrombopag Olamine Tablets (25 mg) in Healthy Chinese Subjects in the Fed State
Brief Title: Bioequivalence Study of Eltrombopag Olamine Tablets in Healthy Subjects in the Fed State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TQZ3469-BE-01
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-01

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: single-dose of test formulation+single-dose of reference formulation (Active Comparator): 18 subjects were enrolled, of whom 9 received the trial drug and 9 received reference preparation.
  Interventions: Drug: Group 1: single-dose of test formulation+single-dose of reference formulation
- Group 2: single-dose of reference formulation+single-dose of test formulation (Active Comparator): 18 subjects were enrolled, of whom 9 received the trial drug and 9 received reference preparation.
  Interventions: Drug: Group 2: single-dose of reference formulation+single-dose of test formulation

INTERVENTIONS:
Drug: Group 1: single-dose of test formulation+single-dose of reference formulation — Eltrombopag olamine is a small molecule non peptide thrombopoietin receptor agonist.
  Arms: Group 1: single-dose of test formulation+single-dose of reference formulation
Drug: Group 2: single-dose of reference formulation+single-dose of test formulation — Eltrombopag olamine is a small molecule non peptide thrombopoietin receptor agonist.
  Arms: Group 2: single-dose of reference formulation+single-dose of test formulation

SUMMARY:
The overall design of this clinical study is a single center, randomized, open label, single dose, two sequence, two cycle bioequivalence trial in healthy individuals under fed conditions. According to the randomized crossover self-control method, healthy volunteer subjects were orally administered with Eltrombopag Olamine Tablets produced by Chia Tai Tianqing Pharmaceutical Group Co., Ltd. Evaluate the human bioequivalence of single dose Reference Listed Drug (RLD) after meals, providing reference for clinical evaluation and medication use.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 to 65 years, inclusive of both 18 and 65 years old;
* Male subjects with a weight of not less than 50.0 kilograms, and female subjects with a weight of not less than 45.0 kilograms; Body Mass Index (BMI) = weight (kg) / height2 (m2), with a BMI range of 18 to 28 kg/m2, inclusive of the boundary values;
* Subjects willing to abstain from childbearing from 2 weeks prior to screening until 6 months after the last administration of the study medication, and voluntarily adopt effective contraceptive measures, with no plans for sperm or egg donation, and ensure the use of one or more non-pharmaceutical contraceptive methods during sexual activity from 2 weeks prior to screening until 6 months after the last administration of the study medication;
* Subjects must sign an informed consent form before the trial, fully understand the content, process, and potential adverse reactions of the trial, and be able to complete the study according to the requirements of the trial protocol.

Exclusion Criteria:

* Subjects with any clinically significant abnormal clinical manifestations that have occurred or are ongoing and require exclusion, including but not limited to neurological/psychiatric, respiratory, cardiovascular, gastrointestinal (any history of gastrointestinal diseases affecting drug absorption), hematopoietic and lymphatic systems, hepatorenal function, endocrine system, and immune system diseases;
* Subjects with any disease that increases the risk of bleeding, such as hemorrhoids, acute gastritis, or gastric and duodenal ulcers, or with any coagulation disorders (such as von Willebrand's disease or hemophilia) or a history of bleeding disorders;
* Subjects with clinically significant abnormalities in physical examination, vital sign measurements, electrocardiogram, and laboratory tests;
* Subjects with clinically significant abnormalities in prothrombin time (PT) and activated partial thromboplastin time (APTT) tests;
* Subjects with abnormal and clinically significant tests for hepatitis B surface antigen, antibodies to hepatitis C virus, antibodies to human immunodeficiency virus, or antibodies to Treponema pallidum;
* Subjects with a history of allergy to eltrombopag or its excipients;
* Subjects who have donated blood or experienced significant blood loss (≥400mL) within three months prior to the trial;
* Subjects with difficulty swallowing tablets;
* Subjects with a history of fainting at the sight of needles or blood, or who cannot tolerate venipuncture;
* Subjects who have taken any medication that alters liver enzyme activity or combined with inhibitors or inducers of CYP3A4, P-gp, or Bcrp, such as itraconazole, ketoconazole, or quinupristin/dalfopristin, within 28 days before the first intake of the study medication;
* Subjects who have taken any prescription or over-the-counter drugs, any vitamin products, or herbal remedies within 28 days before the first intake of the study medication;
* Subjects who have taken the investigational drug or participated in other drug clinical trials and received corresponding study medications within the last three months;
* Subjects with a history of drug abuse within the last six months, or who have used drugs within the last three months, or who test positive for drug abuse screening;
* Subjects with a history of alcohol abuse within the last six months, defined as a weekly alcohol intake exceeding 14 units (1 unit = 360 mL of beer with 5% alcohol content or 45 mL of spirits with 40% alcohol content or 150 mL of wine with 12% alcohol content), or who cannot abstain from alcohol during the trial period;
* Subjects who smoke more than 5 cigarettes per day within the last six months, or who cannot cease using any tobacco products during the trial period;
* Subjects who have consumed any food or drink rich in flavonoids or furanocoumarins, such as grapefruit, pomelo, mango, dragon fruit, grape juice, or orange juice, within 48 hours before administration;
* Subjects who have consumed any food or drink containing caffeine, tea, or xanthine within 48 hours before administration;
* Subjects who have special dietary requirements during the trial period and cannot comply with the provided diet and corresponding regulations;
* Subjects who engage in intense exercise or have significant changes in exercise habits during the trial period;
* Subjects whom the investigator deems unsuitable for enrollment for other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration (Cmax) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72hours after administration
  Maximum Concentration
Time to maximum concentration (Tmax) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72hours after administration
  Time to maximum concentration following drug administration.
Area under the drug-time curve (AUC) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72hours after administration
  Area under the drug-time curve
Apparent terminal elimination half-life (t1/2) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72hours after administration
  Apparent terminal elimination half-life following drug administration
Apparent volume of distribution (Vd/F) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72hours after administration
  Apparent volume of distribution
Clearance rate (CL/F) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72hours after administration
  Clearance rate
Apparent terminal elimination rate constant (λz) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72hours after administration
  Apparent terminal elimination rate constant
Relative bioavailability (F) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72hours after administration
  Relative bioavailability

SECONDARY OUTCOMES:
Incidence of adverse events | From the date of randomization until the date of withdrawal from the clinical trial for any reason, assessed up to 18 days
  Occurrence of all adverse events (aes), serious adverse events (SAEs), and treatment-related adverse events (TEAEs) were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Changchun University of Traditional Chinese Medicine Affiliated Hospital, Changchun, Jilin, China

REFERENCES:
- [Derived] Wu K, Ren Q, Wang Y, Zhou Y, Liu Z, Cheng Y, Deng Q, Cui Y, Yang H. A Single-Center, Randomized, Open-Label, Two-Formulation, Two-Sequence, Two-Period Crossover Study to Evaluate the Bioequivalence of Two Eltrombopag Olamine Tablets (25 mg) in Healthy Chinese Subjects in the Fed State. Clin Drug Investig. 2026 Feb 7. doi: 10.1007/s40261-026-01528-0. Online ahead of print. PMID 41653397